CLINICAL TRIAL: NCT06390241
Title: Avidination for Radionuclide THerapy (A.R.THE.) in Nonpalpable Breast Cancer
Brief Title: Avidination for RadionuclideTHerapy in Nonpalpable Breast Cancer
Acronym: ARTHE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Target enrolment was not met. The trial is terminated because the radiopharmaceutical is not produced under GMP
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.14
Record Dates: First submitted 2024-04-17; First posted 2024-04-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: non-palpable breast lesions; infiltrating breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avidin-biotin-Dota-90Y (Experimental): The total planned enrollment for this study is up to approximately 52 patients for Part 1 (dose-escalation) and Part 2 (dose expansion). Up to 18 patients will be enrolled in Part 1 (depending on dose-escalation) and 40 patients in dose expansion in Part 2. The 6 patients evaluated for dosimetry in Part 1 will also be evaluated in part 2.
  Interventions: Drug: Avidin-biotin-Dota-90Y

INTERVENTIONS:
Drug: Avidin-biotin-Dota-90Y — Within 7-8 days after the VABB procedure, 6-10 mg avidin in 1 ml saline will be administered at the site of the occult carcinoma. Subsequently, 90Y DOTA-biotin in the range of 28-57-126 MBq (3 activity levels investigated) will be injected locally immediately after avidin injection.

SUMMARY:
This is an interventional, open-label, non comparative phase 2 trial enrolling patients with nonpalpable breast cancer

DETAILED DESCRIPTION:
Nonpalpable breast lesions (NPBLs) represent approximately 30% of the overall tumoral breast lesions undergoing surgery. The Vacuum-Assisted Breast Biopsy (VABB) is a device for needle breast biopsy usefully applied in NPBL. The procedure is highly effective for the diagnosis of NPBLs, with minimal negative effects. The specimen volume obtained through this procedure is great enough to replace the diagnostic surgical excisional biopsy and frozen section intraoperative examination. Biopsies obtained through this method sometimes allow the complete excision of the lesion, representing a valid alternative to the excisional biopsy in case of benign lesion less than 15 mm in size.

After VABB procedure about 10-30% of patients have a complete removal of the neoplastic lesion. About 30% of patients are disease free after surgery because the lesion has been totally removed through diagnostic VABB procedure. The rationale of this project is to treat residual microscopic disease through a radionuclide therapy. Our idea is to administer, following VABB procedure, an avidin-biotin-DOTA-90Y (where DOTA stands for 1,4,7,10-tetra-azacyclododecane-N,N',N'',N'''-tetraacetic acid and Y stands for yttrium) compound into the lesion site in order to eliminate residual tumour cells. The ARTHE approach should increase the rate of disease free cases after excisional biopsy.

The primary objective of this open-label phase I trial is to evaluate the safety of avidin-biotin-DOTA-90Y combination in patients with nonpalpable breast cancer undergoing Vacuum-Assisted- Breast- Biopsy (VABB). The co-primary objective is the evaluation of the preliminary anti-tumor activity of the treatment. The secondary objective is to evaluate the dosimetry and biodistribution of avidin-biotin-DOTA-90Y after loco-regional injection under ultrasound guidance.

ARTHE procedure consists of the ultrasound guided injection of Avidin into the breast tissue corresponding to VABB site followed by an injection of Biotin-DOTA-90Y. The injected Biotin-DOTA-90Y will be in a range 28-126 MBq (megabecquerel) (0.2- 0.3 mL, specific activity of 3.7 GBq/mg) (gigabequerel/milligrams). The investigators will inject 6-10 mg of avidin in a volume of 0.3-0.5 mL, followed by biotin-DOTA-90Y immediately after avidin injection.

The hypothesis that a treatment with avidin-biotin-DOTA-90Y is able to destroy residual cancer cells after VABB will be verified by surgery.

The duration of ARTHE procedure is 3 days, including dosimetry evaluation. Patients will receive conservative surgical treatment (4-7 weeks from ARTHE treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have diagnosis of occult breast cancer on the basis of mammography (BIRADS's score 4 - 5)/ultrasound (SCORE 4-5).
2. Pathological diagnosis of in situ or infiltrating breast carcinoma (any histotype)
3. Tumor size >5 and ≤15 mm (at least 13 mm from the skin surface)
4. Female, 18≤age≤75.
5. ECOG (Eastern Cooperative Oncology Group) performance status <2
6. Patients scheduled to receive conservative surgical treatment
7. The effects of investigational medicinal product (IMP) on the developing human fetus are unknown. For this reason and because IMP in this trial is known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion. See Appendix E for the "Recommendations related to contraception and pregnancy testing in clinical trials". Should a woman become pregnant or suspect she is pregnant, she should inform her treating physician immediately.
8. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Histotype different from carcinoma
2. Paget carcinoma
3. Lesions located near to axilla region or skin <13 mm
4. Ongoing pregnancy or breastfeeding
5. Previous treatment with avidin
6. Referred allergy to eggs or latex
7. Patients with metastases should be excluded from this clinical trial.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Patients with previous radiotherapy and/or operation on the same breast, with diffuse microcalcifications will be excluded.
10. Patients with known BRCA (BReast CAncer gene), PALB2 (Partner and Localizer of BRCA2) and CHECK2 (Checkpoint Kinase 2) mutations, grade 3 risk profile or indication to perform a test for germline mutations based on disease characteristics
11. Multifocal tumors are not eligible for the study.
12. History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS (overall survival) rate >90%).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Safety of avidin-biotin-Dota-90Y | 4-7 weeks
  The primary endpoint is the local toxicity evaluated according to Radiation Therapy Oncology Group (RTOG) scale. According to the RTOG scale grades range from 0 to 5, where 0 represents no change over baseline and 5 represents any toxicity which causes death.
Safety of avidin-biotin-Dota-90Y | 4-7 weeks
  The primary endpoint is the systemic toxicity evaluated according to NCI-CTCAE (The U.S. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events) Version 5.0
Anti-tumor activity of avidin-biotin-Dota-90Y | 4-7 weeks
  The co-primary endpoint is the evaluation of the complete pathological response rate, defined as the absence of residual invasive and in situ cancer or DCIS (ductal carcinoma in situ), on hematoxylin and eosin evaluation of the complete resected breast specimen and of all sampled regional lymph nodes (i.e., ypT0 ypN0 in the current AJCC staging system).

SECONDARY OUTCOMES:
Dose-response | 48-72 hours after injection
  Serial PET (positron emission computed tomography)/CT (computerized tomography) scan will be performed at defined time intervals after radiopharmaceutical administration. The number of PET/CT scans depends on the presence of wash-out documented by the whole body image acquired with SPECT/CT scanner. A dedicated software will be used to segment the region of interest, to quantify the activity inside the target region, and to estimate the number of disintegrations, that is the input data for absorbed dose calculation. For the tumor absorbed dose calculation, the spherical volume approximation is used with a uniform activity distribution. The tumor mass is estimated from the CT scan.
  From the computed data, a detailed report relative to absorbed dose to the tumor and neighboring organs treated with avidin-biotin-DOTA-90Y will be prepared, in order to provide a dose-response relationship for toxicity avoidance.
Biodistribution | 1-3 hours after injection
  The whole-body image will be used to evaluate 90Y biodistribution in the body and to verify that the injected activity is really localized in the breast tissue. In this case, the treatment can be considered as locoregional, with the uptake concentrated in a limited region of the breast, without the involvement of other organs. To evaluate the assumption of a localized uptake in the tumor lesion, the patients will undergo just one PET/ CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Matteucci, Principal Investigator — IRCCS IRST
Locations (1):
- IRCCS Istituto ROmagnolo per lo Studio dei Tumori "Dino Amadori"-IRST S.r.l., Meldola, Forlì Cesena, Italy

IPD SHARING:
Plan to Share IPD: No